CLINICAL TRIAL: NCT06641622
Title: Study of the Correlation Between Donor CIRBP and Transplanted Kidney Function
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qianghua Leng, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: II-2024-046-02
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplant; Complications; Delayed Graft Function
Keywords: kidney transplantation; cold-inducible RNA binding protein; delayed graft function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- delayed graft function: DGF was defined as a decrease in daily plasma creatinine of less than 10% from the previous day for 3 consecutive days within 1 week postoperatively, or if serum creatinine (SCr) did not decrease to 400 μmol/L within 1 week after surgery
  Interventions: Diagnostic Test: Prediction of delayed graft function
- immediate graft function: Recipients who did not develop DGF were categorized as IGF

INTERVENTIONS:
Diagnostic Test: Prediction of delayed graft function — Donor plasma CIRBP levels were measured using an ELISA kit to evaluate their association with DGF incidence
  Groups: delayed graft function

SUMMARY:
Deceased donors and recipients who successfully completed kidney transplantation between 2016 and 2019 were included in this study. Donor plasma CIRBP levels were measured using an ELISA kit to evaluate their association with DGF incidence.

DETAILED DESCRIPTION:
The study was a retrospective open cohort study that included deceased patients from January 2016 to December 2019. It adhered to the guidelines of the National Program for Deceased Organ Donation in China and involved successful kidney donors from the Third Affiliated Hospital of Sun Yat-sen University. Donors were excluded if they met any of the following conditions: (a) lacked a blood specimen; (b) had contaminated blood specimens affecting CIRBP levels; (c) were recipients who underwent combined multi-organ transplants; (d) were participating in other clinical trials; (e) had a history of organ transplantation; (f) had other conditions deemed unsuitable for enrollment by the investigator. Blood specimens were collected from donors by Organ Procurement Organizations (OPOs) and used for various studies with the donors' consent. All recipients (207 recipients, 207 donors) were followed up in the long term after transplantation.

The investigators followed the principles outlined in the Declaration of Helsinki (20) and the Declaration of Istanbul . Approval for this study was obtained from the Human Organ Transplantation and Ethics Committee of Sun Yat-sen University. The Ethics Committee was formed in compliance with the World Health Organization's Operational Guidelines for Ethics Committee Review of Biomedical Research. Organ allocation was performed in a fair and transparent manner via the Chinese Organ Transplant Response System. The type of donation was voluntarily determined by the donor's family, and the recipient underwent follow-up after transplantation. Both the donor's family and the recipient provided consent for the use of samples and clinical data in research.

Donor data were obtained from the China Organ Transplant Response System, completed by members of organ transplant organizations. Additionally, some donor information was supplemented from clinical electronic medical records. Recipient data were derived from clinical electronic records alone. Investigators categorized donors and recipients into delayed graft function (DGF) and immediate graft function (IGF) groups based on the recipient's early renal function status. DGF was defined as a decrease in daily plasma creatinine of less than 10% from the previous day for 3 consecutive days within 1 week postoperatively, or if serum creatinine (SCr) did not decrease to 400 μmol/L within 1 week after surgery. Recipients who did not develop DGF were categorized as IGF. Primary nonfunction (PNF) was diagnosed in patients requiring continuous dialysis after surgery or retransplantation. Additionally, expended criteria donors were defined as those aged over 60 years, or between 50 and 59 years meeting at least two of the following criteria: final serum creatinine > 133 μmol/L, cerebrovascular accident as the cause of death, and a history of hypertension.

Sample Collection Whole blood specimens were obtained from the donor in the operating theater before organ retrieval and transported on crushed ice to the laboratory, with an average transit duration of 2 hours. For serum preparation, the whole blood specimens were left at room temperature for 2 hours, then centrifuged at 1000 g for 15 minutes at a temperature of 2-8°C. The resulting supernatant was collected and stored at -80°C within the laboratory. Before testing, the serum samples were thawed on crushed ice and centrifuged again at 1000 g for 15 minutes at 2-8°C.

Measurement Of Cold Inducible RNA Binding Protein Level Serum CIRBP was detected using an ELISA kit (CSB-EL005440HU). The protein standard was diluted according to the instructions, and 100 µl of different concentrations of standard and samples (1:10 dilution) were added to a 96-well plate in duplicate. The plate was incubated at 37°C for 2 hours in the dark. Following incubation, the liquid in the wells was discarded, and 100 µl of biotin-labeled antibody working solution was added to each well. After incubating at 37°C for 1 hour, the plate was washed three times with washing solution. Subsequently, 100 µl of horseradish peroxidase-labeled affinity solution was added to each well. After an additional 1-hour incubation at 37°C, the plate was washed five times. Then, 90 µl of substrate solution was added to each well, and after a 15-minute color development at 37°C, 50 µl of termination solution was used to stop the reaction. The absorbance was measured at 450 nm within 5 minutes using a microplate reader, and concentrations were calculated based on the standard curve.

ELIGIBILITY:
Inclusion Criteria:

* Kidney donors who meet the criteria for donation;
* First-time kidney transplant recipients;
* Transplantation using cadaveric donor kidneys;
* Signing of the Human Organ Donation Relative Acknowledgement Registration Form.

Exclusion Criteria:

* those without a blood specimen;
* contamination of the blood specimen affecting the CIRBP level;
* recipients of combined multi-organ transplants;
* those participating in other clinical trials;
* the existence of a previous history of other organ transplants;
* any other condition that, in the opinion of the investigator, makes enrolment unsuitable.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our study was a retrospective open cohort study that included deceased patients from January 2016 to December 2019. It adhered to the guidelines of the National Program for Deceased Organ Donation in China and involved successful kidney donors from the Third Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
recipients developed delayed graft function | within 1 week after surgery
  DGF was defined as a decrease in daily plasma creatinine of less than 10% from the previous day for 3 consecutive days within 1 week postoperatively, or if serum creatinine (SCr) did not decrease to 400 μmol/L within 1 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qianghua Leng, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Share the data on Public management platform for clinical trials ResMan
Supporting Information: Study Protocol, SAP, CSR
Time Frame: March 2025, for 3 years

REFERENCES:
- [Background] Yang R, Zhan M, Nalabothula NR, Yang Q, Indig FE, Carrier F. Functional significance for a heterogenous ribonucleoprotein A18 signature RNA motif in the 3'-untranslated region of ataxia telangiectasia mutated and Rad3-related (ATR) transcript. J Biol Chem. 2010 Mar 19;285(12):8887-93. doi: 10.1074/jbc.M109.013128. Epub 2010 Jan 26. PMID 20103595
- [Derived] Leng Q, Ma M, Tang Z, Jiang W, Han F, Huang Z. Assessing donor kidney function: the role of CIRBP in predicting delayed graft function post-transplant. Front Immunol. 2025 Jan 17;15:1518279. doi: 10.3389/fimmu.2024.1518279. eCollection 2024. PMID 39896811